CLINICAL TRIAL: NCT06766201
Title: Effect of Use of Calcium Hydroxide and Metformin as Intracanal Dressings in Healing of Apical Periodontitis in Mature Permanent Mandibular Molars: A Randomized Clinical Trial
Brief Title: Effect of Use of Calcium Hydroxide and Metformin Intracanal Medicament After NSRCT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Principal Investigator, Sanjay Tewari, Principal, Postgraduate Institute of Dental Sciences Rohtak
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMBIKA TEKTA
Record Dates: First submitted 2024-06-04; First posted 2025-01-09 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Apical Periodontitis
Keywords: AP, metformin, calcium hydroxide, medicament
MeSH Terms: conditions — Periapical Periodontitis | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calcium hydroxide group (No Intervention): Calcium hydroxide is mixed with propylene glycol
- metformin group (Experimental): metformin mixed with propylene glycol
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin mixed with propylene glycol
  Other Names: MF
  Arms: metformin group

SUMMARY:
Goal of this randomized clinical trial is evaluate the effect of Calcium Hydroxide and Metformin Intracanal Medicament on periapical healing after NSRCT. Population includes systemically healthy patient with radiographic evidence of apical periodontitis PAI score more then 3 will be recruited . Outcome will be assessed using periapical index scoring system at 6 and 12 months follow up period.

DETAILED DESCRIPTION:
AIM: To compare the efficacy of calcium hydroxide and metformin intracanal medicaments in healing of apical periodontitis in mature permanent mandibular molars. Objectives Primary objective: To determine the effect of calcium hydroxide and metformin intracanal medicaments on healing of apical periodontitis in mature permanent mandibular molars using periapical index (PAI) score. Secondary objective: assess postoperative pain after chemo mechanical preparation and intracanal dressing of calcium hydroxide or metformin using visual analogue scale (VAS)

Clinical procedure Mature permanent mandibular teeth with diagnosis of apical periodontitis (as confirmed clinically & by periapical radiograph) will be chosen for the study. 17 Patients will be randomly allocated to either of the two groups- Group A (calcium hydroxide), Group B (Metformin). The tooth will be anesthetized using 2% lidocaine with 1:100000 adrenaline followed by rubber dam isolation. Caries excavation will be done and access cavity will be made. Coronal flaring & enlargement will be performed with rotary NiTi orifice enlargers to obtain straight -line access to the apical third of each root. Hand files No. 10, 15 and 20 will be used till working length (WL) to prepare a smooth reproducible glide path Working length will be obtained with the help of electronic apex locator (Root ZX) and confirmed radiographically. Canals will be then prepared using the Crown down technique with rotary instruments.

5ml of 5.25% sodium hypochlorite is used as irrigate after each instrument. After completion of canal instrumentation, all canal will be irrigated with 17% ethylenediamine-tetra acetic acid for 1 minute followed by a final irrigation with 5.0 ml of 5.25% sodium hypochlorite. Patency will maintained by placing a 10 k file 1 mm beyond the apical foramen after each instrument change. Canals will be dried with absorbent paper points and filled with a Calcium hydroxide with propylene glycol in control group A and will be filled with 1% Metformin with propylene glycol in control group B .Both paste will be paced in canal by lentulospiral and the access cavity restored with intermediate restorative material (IRM). The patient will be recalled after 1 week and evaluated for post operative pain.

At the next appointment, the paste will be removed with H- files and copious irrigation with 5.25% NaOCl; and dried with paper points. Canals will be obturated with the Gutta Percha and Zinc Oxide- Eugenol based sealer.

After obturation, the cavity will be restored . Immediate postoperative radiograph will then be taken. Follow up clinical and radiographic examinations will be carried out at 6 month & 12 month period.

ELIGIBILITY:
Inclusion Criteria:

1. Mature permanent mandibular molar with necrotic pulp (absence of response to cold and electric pulp tester) and apical periodontitis requiring primary root canal treatment with radiographic evidence of periapical radiolucency (periapical index score ≥ 3).
2. Age - Above 18 years
3. Non-contributory medical history (ASA 1)
4. Periodontally healthy tooth (probing depth <4mm)

Exclusion Criteria:

1. Patients who do not provide authorization for participation in the study
2. History of analgesic intake in the previous 1 week, or antibiotic intake in 1 month
3. Mandibular molar with no opposing teeth.
4. Patients whose tooth had been previously accessed or endodontically treated.
5. Patient on systemic MF or medication that interfere periapical healing
6. Presence of bleeding on opening of pulp chamber.
7. Diabetic, immunocompromised and pregnant patient.
8. Teeth with cracks, fracture, internal and external resorption.
9. Any medications that alter bone metabolism such as, immunosuppressive drugs, corticosteroids, hormone replacement therapy ,selective serotonin reuptake inhibitors, intravenous bisphosphonates, and/or antiresorptive treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
periapical healing using the Periapical index score | 6 and12 months follow .
  clinical and radiographic healing clinical and radiographic success at 6 and12 months follow .

SECONDARY OUTCOMES:
Clinical success | 6 and12 months follow .
  Absence of pain and tenderness to percussion/palpation, the absence of sinus or any associated soft-tissue swelling, tooth mobility of grade 1 or less, and no deterioration in periodontal probing depth as compared with baseline measurements

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sanjay Tewari, MDS, Study Director — Post Graduate Institute Of Dental Sciences,Rohtak
Locations (1):
- Ambika Tekta, Rohtak, Haryana, India